CLINICAL TRIAL: NCT02977572
Title: Non-Invasive Mechanical Ventilation Versus Continuous Positive Airway Pressure Relating to Cardiogenic Pulmonary Edema in an Intensive Care Unit
Brief Title: Non-invasive Ventilation Versus Continuous Positive Airway Pressure in Cardiogenic Pulmonary Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Castellón (Other)
Responsible Party: Principal Investigator, ALBERTO BELENGUER MUNCHARAZ, MD, Phd, INTENSIVE CARE UNIT, Hospital General Universitario de Castellón
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGU Castellon-002
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Cardiogenic Pulmonary Oedema
Keywords: Non-invasive ventilation,; continuous positive airway pressure; cardiogenic pulmonary oedema,; acute respiratory failure
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Invasive ventilation (NIV group) (Experimental): For the NIV group, a BiPAP Vision was used, by setting the Inspiratory Positive Airway Pressure (IPAP) at a level that was required to achieve a tidal volume of approximately 8-10 ml/kg. Also an Expiratory Positive Airway Pressure (EPAP) was set at a minimum of 5 cmH20 during the first hour, gradually increasing until there was a clinical improvement. Fraction inspiratory of oxygen (FiO2) was applied to maintain a transcutaneous arterial oxygen saturation (SaO2) of 92%-94%. NIV was continuously applied until there was a clinical and/or a gasometrical improvement, at which time they were replaced by a Venturi mask with FiO2 of 0.4.
  Interventions: Device: Non-Invasive Ventilation
- Continuous Positive AirwayPressure CPAP (Placebo Comparator): The CPAP was applied by using a flow generator with adjustable fractional inspired oxygen (FiO2). This was connected to the Positive End-Expiratory Pressure (PEEP) valve that was placed in the face mask. In the second instance, the CPAP system that was used was a Boussignac CPAP System Flow Jet. The Boussignac valve takes gas from a single source and splits it in order to create four high flow jets. These jets converge in the chamber creating a virtual valve. A initial level of 5cmH20 of PEEP was recommended for the first hour of ventilation, with subsequent increments (up to 15cmH20) until a clinical improvement was obtained. CPAP was continuously applied until there was a clinical and/or a gasometrical improvement, at which time it was replaced by a Venturi mask.
  Interventions: Device: Continuous Positive AirwayPressure CPAP

INTERVENTIONS:
Device: Non-Invasive Ventilation — In arm description
  Arms: Non-Invasive ventilation (NIV group)
Device: Continuous Positive AirwayPressure CPAP — In arm description
  Arms: Continuous Positive AirwayPressure CPAP

SUMMARY:
The aim of the present study was to demonstrate that an Non-Invasive Ventilation (NIV) performs better than a Continuous Positive Airway Pressure (CPAP) in the management of Cardiogenic Pulmonary Edema (CPE) within an Intensive Care Unit (ICU) setting.

DETAILED DESCRIPTION:
Continuous Positive Airway Pressure (CPAP) and Non-Invasive Ventilation (NIV), has played a decisive role in the treatment of Acute Respiratory Failure (ARF) secondary to Cardiogenic Pulmonary Edema (CPE). The use of either CPAP or NIV has resulted in greater clinical improvements than the ones that have been previously obtained by using a standard medical therapy. Although there is a strong indication for NIV in hypercapnic patients, the situation whether NIV is superior to CPAP remains unclear, and hence, both have been recommended.

NIV and CPAP have both been successfully used in patients admitted to an Intensive Care Unit (ICU) suffering from CPE. However, few trials have been published on the ICU scenario. In addition, Acute Coronary Syndrome (ACS) has been considered to be an exclusion criterion in several trials.

At the time of the onset of CPE, either in the Emergency Department (ED) or in the ward, all participants received a standard medical therapy (oxygen through a Venturi mask, morphine, intravenous nitroglycerin if their systolic blood pressure >160 mmHg, together with loop diuretics), all at the discretion of the attending physician. In the absence of a clinical improvement [dyspnea, respiratory rate >25rpm, transcutaneous arterial oxygen saturation (SaO2) <90%], the participant was admitted to the ICU and assigned to the NIV group or the CPAP group, regardless of the treatment that they had received in the ED. The participants that were admitted to the ICU at the onset of CPE were randomised without a trial of medical treatment. The assignment of each group was performed by opening a sealed envelope following a prior randomisation by using a computerised system.

Statistical. A comparative analysis was conducted by using the Student's t-test or the Mann-Whitney test for a comparison of the quantitative variables for the parametric and non-parametric characteristics, respectively. For the qualitative variables, the investigators used the Chi-Square statistic or Fisher's exact test. A statistical significance was reached if P<0.05. The cumulative probability of survival was compared by using a Kaplan-Meier estimation of survival and a Log-Rank Test to compare both of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants suffering from CPE, defined as having the presence of dyspnea, respiratory rate >25 breaths/minute, the use of accessory respiratory muscles, cyanosis, cold sweats, bilateral crackles and/or wheezing on pulmonary auscultation, hypoxaemia, hypertension, and a predominance of bilateral pulmonary infiltrates upon a chest radiography (if available).
* The potential causes of CPE have been understood to be Acute Coronary Syndrome (ACS) with or without a persistent ST-segment elevation, hypertensive emergency, valvulopathy, acute arrhythmia, endocarditis, or decompensation due to a chronic heart failure.

Exclusion Criteria:

* The exclusion criteria were: a refused consent, the patient's inability to cooperate, severe encephalopathy (Glasgow Coma Score <10)
* Anatomical difficulty when adjusting the face mask, non-cardiogenic Acute Respiratory Failure (pneumonia, blunt chest trauma, or chronic obstructive pulmonary disease)
* Respiratory or cardiac arrest on admission, together with the need for an immediate intubation.
* Specific cardiac contraindications were also considered, including: cardiogenic shock on admission established by systolic blood pressure (SBP) <90 mmHg, or a dependence on vasoactive drugs (norepinephrine >0.5 µg/kg/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALBERTO BELENGUER-MUNCHARAZ, MD, Principal Investigator — INTENSIVE CARE UNIT. HOSPITAL GENERAL CASTELLO

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Invasive Ventilation (NIV Group): For the Non-Invasive ventilation group, a BiPAP Vision was used, by setting the Inspiratory Positive Airway Pressure (IPAP) at a level that was required to achieve a tidal volume of approximately 8-10 ml/kg. Also an Expiratory Positive Airway Pressure (EPAP) was set at a minimum of 5 cmH20 during the first hour, gradually increasing until there was a clinical improvement. Fraction inspiratory of oxygen (FiO2) was applied to maintain a transcutaneous arterial oxygen saturation (SaO2) of 92%-94%. NIV was continuously applied until there was a clinical and/or a gasometrical improvement, at which time they were replaced by a Venturi mask with FiO2 of 0.4.
  Non-Invasive Ventilation: In arm description
- Continuous Positive Airway Pressure (CPAP) Group: The Continuous Positive Airway Pressure was applied by using a flow generator that was capable of delivering a flow of 140 Liter/minute, with adjustable fractional inspired oxygen that ranged from 0.3 to 1.0. This was connected to the Positive End-Expiratory Pressure valve that was placed in the face mask. In the second instance, the CPAP system that was used was a Boussignac CPAP System. The Boussignac valve takes gas from a single source and splits it in order to create four high flow jets. These jets converge in the chamber creating a turbulence which creates a virtual valve. A minimal initial level of 5cmH20 of PEEP was recommended for the first hour of the CPAP, with subsequent increments (up to 15cmH20) until a clinical improvement was obtained. CPAP was continuously applied until there was a clinical and/or a gasometrical improvement, at which time they were replaced by a Venturi mask with FiO2 of 0.4.
  Continuous Positive Airway Pressure: In arm description
Period: Overall Study
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Started | 58 | 56
Completed | 56 | 54
Not Completed | 2 | 2
Not completed — Exclusion criterion | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Continuous Positive Airway Pressure (CPAP) Group: The CPAP was applied by using a flow generator that was capable of delivering a flow of 140 Liter /minute, with adjustable fractional inspired oxygen (FiO2) that ranged from 0.3 to 1.0. This was connected to the Positive End-Expiratory Pressure (PEEP) valve that was placed in the face mask. In the second instance, the CPAP system that was used was a Boussignac CPAP System Flow Jet. The Boussignac valve takes gas from a single source and splits it in order to create four high flow jets. These jets converge in the chamber creating a turbulence which creates a virtual valve. A minimal initial level of 5cmH20 of PEEP was recommended for the first hour of the CPAP, with subsequent increments (up to 15cmH20) until a clinical improvement was obtained. CPAP was continuously applied until there was a clinical and/or a gasometrical improvement, at which time they were replaced by a Venturi mask with FiO2 of 0.4.
  Continuous Positive Airway Pressure: In arm description
- Total: Total of all reporting groups
Arm/Group | Continuous Positive Airway Pressure (CPAP) Group | Non-Invasive Ventilation (NIV Group) | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 40 | 38 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 35 | 42 | 77

OUTCOME MEASURES:

1. Primary Outcome: Need for an Endotracheal Intubation Within Seven Days After Onset of Cardiopulmonary Edema at the Intensive Care Unit
Time Frame: Whitin seven days after onset of cardiopulmonary edema at the Intensive Care Unit
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
Participants | 5 | 5
Statistical Analysis 1: Comparison: Non-Invasive Ventilation (NIV Group) vs Continuous Positive Airway Pressure (CPAP) Group; Based upon previous results, the investigators considered that the need for an intubation could be reduced by 15% [19% in the CPAP group (control) vs. 4% in the NIV group (study)]. The estimated sample size was 55 participants in each group (confidence interval [1-α] = 90% and power [1-β] = 85%); Test type: Superiority or Other; p = 1.000, Chi-squared

2. Secondary Outcome: Duration of the Ventilation
Description: Period of ventilation (either noninvasive ventilation or continouos positive airway pressure) while the patient suffers from acute respiratory failure secondary to cardiopulmonary edema
Time Frame: Time (hours) from start of ventilation until the removal of both devices because of improve or failure
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
hours | 16 [6 to 34] | 10 [2 to 31]

3. Secondary Outcome: Ventilator Acquired Pneumonia
Description: Pulmonary infections (%) during stay at intensive care unit
Time Frame: Pulmonary infection at intensive care unit diagnosed until 72 hours after removal of ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Positive Airway Pressure (CPAP) Group | Non-Invasive Ventilation (NIV Group)
Number analyzed (Participants) | 56 | 54
Participants | 3 | 1

4. Secondary Outcome: Acute Renal Failure
Description: Development of acute renal failure measured as increase of level of creatinine
Time Frame: Acute Renal Failure during intensive care unit stay (at discharge from intensive care unit)
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
Participants | 12 | 13

5. Secondary Outcome: Length of Stay at Intensive Care Unit
Description: Length of stay of the patient at Intensive Care Unit
Time Frame: Length of stay (days) at Intensive Care Unit at discharge from intensive care unit.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
days | 3 [2 to 6] | 4 [1 to 7]

6. Secondary Outcome: Length of Hospital Stay
Description: All the time (days) the patient stays at the hospital
Time Frame: Length of stay (days) at hospital at discharge from hospital
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
days | 12 [7 to 17] | 14 [6 to 24]

7. Secondary Outcome: Intensive Care Unit Mortality
Description: Mortality (%) at Intensive Care Unit
Time Frame: Mortality (%) at Intensive Care Unit at discharge from intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
Participants | 12 | 14

8. Secondary Outcome: 28th Day Mortality
Description: Mortility of patients within of the first 28 days after randomization (either at intensive car unit or at hospital)
Time Frame: Mortality within 28 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
Participants | 13 | 16

9. Secondary Outcome: Hospital Mortality
Description: Mortality during hospital stay (including at Intensive care mortality)
Time Frame: Mortality (%) at Hospital at discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
Number analyzed (Participants) | 56 | 54
Participants | 15 | 17

ADVERSE EVENTS:
Description: Serious and Other Adverse Events were not assessed.
Arm/Group | Non-Invasive Ventilation (NIV Group) | Continuous Positive Airway Pressure (CPAP) Group
All-Cause Mortality (participants affected / at risk) | 15/56 | 17/54
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes